CLINICAL TRIAL: NCT05841160
Title: A Randomized, Double-Blind, Placebo- and Positive Controlled, Crossover, Thorough QT/QTc Study to Evaluate the Effects of a Therapeutic and Supratherapeutic Dose of Ecopipam (EBS-101) on Cardiac Repolarization in Healthy Subjects
Brief Title: Thorough QT/QTc Study to Evaluate the Effects of Ecopipam (EBS-101) on Cardiac Repolarization
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emalex Biosciences Inc. (Industry)
Collaborators: PPD Development, LP (Industry); Clario (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EBS-101-HV-105
Record Dates: First submitted 2023-04-10; First posted 2023-05-03 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: QT/QTc
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 200 mg ecopipam HCL (Experimental): Single 200 mg dose of ecopipam HCL given as 2 x 100 mg ecopipam HCL oral tablets and 4 placebo oral tablets
  Interventions: Drug: Ecopipam Hydrochloride; Drug: Placebo
- 600 mg ecopipam HCL (Experimental): Single 600 mg dose of ecopipam HCL given as 6 x 100 mg ecopipam HCL oral tablets
  Interventions: Drug: Ecopipam Hydrochloride
- 400 mg moxifloxacin (Active Comparator): Single 400 mg dose of moxifloxacin given as 1 x 400 mg oral tablet
  Interventions: Drug: Moxifloxacin
- Placebo (Placebo Comparator): Single oral dose of 6 x placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ecopipam Hydrochloride — oral tablets
  Arms: 200 mg ecopipam HCL; 600 mg ecopipam HCL
Drug: Moxifloxacin — oral tablet
  Arms: 400 mg moxifloxacin
Drug: Placebo — oral tablet
  Arms: 200 mg ecopipam HCL; Placebo

SUMMARY:
THOROUGH QT/QTc STUDY TO EVALUATE THE EFFECTS OF ECOPIPAM (EBS-101) ON CARDIAC REPOLARIZATION

DETAILED DESCRIPTION:
This is a single-center, randomized, partially double-blind (open-label moxifloxacin), placebo- and positive-controlled, 4-way crossover study in healthy subjects. Following a 28 day screening period, eligible subjects will enter the clinical research unit (CRU) on Day -1. A total of 32 subjects will be randomized in a 1:1:1:1 ratio to 1 of 4 treatment sequences (8 subjects per treatment sequence). Subjects will receive the assigned study drug as a single oral dose in the morning on Day 1 of each treatment period (Day 1 [Period 1], Day 8 [Period 2], Day 15 [Period 3], and Day 22 [Period 4]) after an overnight fast. Subjects will have serially matched blood samples (for determination of plasma concentrations) and 12-lead ECGs collected at predose and up to 48 hours after each dose for C QTc analysis. Subjects will be discharged from the CRU 96 hours after the last dose of the study drug (Day 26). A follow-up telephone call will occur 5 ±2 days after discharge (Day 31 ±2).

ELIGIBILITY:
Inclusion Criteria:

* Male or female of nonchildbearing potential
* 18 to 55 years of age
* BMI of 18 to 30 kg/m2, and weight of at least 50 kg for males and 45 kg for females.
* Subject considered by the investigator to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead ECG results, and PE findings.
* Male subjects with female partners of childbearing potential must agree to use a double-barrier method of contraception during the study and agree to continue the use of male contraception for at least 90 days after the last dose of study drug.
* Male subjects must be willing to refrain from donating sperm during study participation and for 90 days after the last dose of study drug.
* The subject is able to provide written informed consent and agrees to comply with all protocol requirements.

Exclusion Criteria:

* Female subjects of childbearing potential or who are currently pregnant or lactating
* Subjects with a history of significant medical illness
* Clinically significant abnormalities on screening tests/exams
* History of or serious risk of committing suicide
* Donation of plasma within 7 days prior to dosing
* Donation of significant loss of blood within 30 days prior to dosing
* Major surgery within 3 months or minor surgery within 1 month prior to CRU admission
* Use of prohibited prescription, over-the-counter medications or natural health products
* Alcohol-based products within 24 hours prior to check-in on Day -1
* Vaccinations within 72 hours prior to check-in on Day -1
* Subjects with a history of any clinically significant ECG or vital sign abnormalities or presence of any clinically significant ECG or vital sign abnormalities or changes at screening or on Day -1
* Positive test result for drugs of abuse, alcohol, or cotinine
* Use of nicotine or nicotine-containing products within 90 days before the first dose of study drug.
* Subjects with a history of excessive alcohol intake or abuse or drug addiction within the last year
* Subjects with a history of allergy, allergic skin rash, asthma, or an intolerance, sensitivity, or photosensitivity to moxifloxacin or ecopipam
* Subjects who have participated in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dose or administration of a biological product in the context of a clinical research study within 90 days prior to the first dose
* Subjects with prior exposure to ecopipam
* Any subject who, in the opinion of the investigator, is not a suitable candidate for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-05-07 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Evaluate ecopipam's effect on the QTc interval after administration of therapeutic and supratherapeutic doses, compared to placebo as a negative control using C-QTc analysis. | Up to Day 25
  ECGs and PK samples will be collected for up to 96 hours after each dose

SECONDARY OUTCOMES:
Evaluate the effect of ecopipam at a therapeutic dose on heart rate | Up to Day 25
  ECGs will be collected for up to 48 hours after each dose
Evaluate the effect of ecopipam at a therapeutic dose on PR interval | Up to Day 25
  ECGs will be collected for up to 48 hours after each dose
Evaluate the effect of ecopipam at a therapeutic dose on QRS interval | Up to Day 25
  ECGs will be collected for up to 48 hours after each dose
Evaluate the effect of ecopipam at a therapeutic dose on T-wave morphology | Up to Day 25
  ECGs will be collected for up to 48 hours after each dose
Evaluate the effect of ecopipam at a therapeutic dose on U wave presence | Up to Day 25
  ECGs will be collected for up to 48 hours after each dose
Evaluate the effect of ecopipam at supratherapeutic dose on heart rate | Up to Day 25
  ECGs will be collected for up to 48 hours after each dose
Evaluate the effect of ecopipam at supratherapeutic dose on PR interval | Up to Day 25
  ECGs will be collected for up to 48 hours after each dose
Evaluate the effect of ecopipam at supratherapeutic dose on QRS interval | Up to Day 25
  ECGs will be collected for up to 48 hours after each dose
Evaluate the effect of ecopipam at supratherapeutic dose on T-wave morphology | Up to Day 25
  ECGs will be collected for up to 48 hours after each dose
Evaluate the effect of ecopipam at supratherapeutic dose on U wave presence | Up to Day 25
  ECGs will be collected for up to 48 hours after each dose
Evaluate the ECG assay sensitivity to detect a change in the QT interval corrected for heart rate using Fridericia's formula (QTcF interval) using 400 mg moxifloxacin as the positive control | Up to Day 25
  ECGs will be collected for up to 48 hours after each dose
Evaluate the effects of ecopipam on the emergence of arrhythmias | Up to Day 25
  ECGs will be collected for up to 48 hours after each dose
Describe the incidence of treatment-emergent adverse events after a single therapeutic dose of ecopipam | Up to Day 33
  AEs will be collected throughout the duration of the study
Describe the incidence of treatment-emergent adverse events after a single supratherapeutic dose of ecopipam | Up to Day 33
  AEs will be collected throughout the duration of the study
Describe the incidence of treatment-emergent adverse events after a single dose of moxifloxacin 400 mg | Up to Day 33
  AEs will be collected throughout the duration of the study
Describe the Cmax of ecopipam after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the Tmax of ecopipam after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUClast of ecopipam after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUCinf of ecopipam after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUCext of ecopipam after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the λz of ecopipam after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the t1/2 of ecopipam after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the Cmax of ecopipam after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the Tmax of ecopipam after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUClast of ecopipam after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUCinf of ecopipam after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUCext of ecopipam after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the λz of ecopipam after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the t1/2 of ecopipam after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the Cmax of EBS-101-40853 after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the Tmax of EBS-101-40853 after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUClast of EBS-101-40853 after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUCinf of EBS-101-40853 after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUCext of EBS-101-40853 after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the λz of EBS-101-40853 after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the t1/2 of EBS-101-40853 after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the Cmax of EBS-101-40853 after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the Tmax of EBS-101-40853 after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUClast of EBS-101-40853 after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUCinf of EBS-101-40853 after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUCext of EBS-101-40853 after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the λz of EBS-101-40853 after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the t1/2 of EBS-101-40853 after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the Cmax of ecopipam glucuronide after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the Tmax of ecopipam glucuronide after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUClast of ecopipam glucuronide after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUCinf of ecopipam glucuronide after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUCext of ecopipam glucuronide after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the λz of ecopipam glucuronide after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the t1/2 of ecopipam glucuronide after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the Cmax of ecopipam glucuronide after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the Tmax of ecopipam glucuronide after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUClast of ecopipam glucuronide after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUCinf of ecopipam glucuronide after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUCext of ecopipam glucuronide after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the λz of ecopipam glucuronide after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the t1/2 of ecopipam glucuronide after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the Cmax of EBS-101-40853 glucuronide after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the Tmax of EBS-101-40853 glucuronide after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUClast of EBS-101-40853 glucuronide after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUCinf of EBS-101-40853 glucuronide after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUCext of EBS-101-40853 glucuronide after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the λz of EBS-101-40853 glucuronide after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the t1/2 of EBS-101-40853 glucuronide after single therapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the Cmax of EBS-101-40853 glucuronide after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the Tmax of EBS-101-40853 glucuronide after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUClast of EBS-101-40853 glucuronide after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUCinf of EBS-101-40853 glucuronide after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUCext of EBS-101-40853 glucuronide after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the λz of EBS-101-40853 glucuronide after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the t1/2 of EBS-101-40853 glucuronide after single supratherapeutic dose of ecopipam | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the Cmax of moxifloxacin after a single dose of moxifloxacin 400 mg | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the Tmax of moxifloxacin after a single dose of moxifloxacin 400 mg | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUClast of moxifloxacin after a single dose of moxifloxacin 400 mg | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUCinf of moxifloxacin after a single dose of moxifloxacin 400 mg | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the AUCext of moxifloxacin after a single dose of moxifloxacin 400 mg | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the λz of moxifloxacin after a single dose of moxifloxacin 400 mg | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis
Describe the t1/2 of moxifloxacin after a single dose of moxifloxacin 400 mg | Up to Day 33
  17 blood samples will be collected at the indicated timepoints for pharmacokinetic analysis

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Austin Phase 1 Clinical Research Unit, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No